CLINICAL TRIAL: NCT03109964
Title: The Affect of Hemostasis With Bipolar Coagulation Versus SURGIFLO Placement on Ovarian Reserve and Future Fertility
Brief Title: The Affect of Hemostasis Technique During Laparoscopic Ovarian Cystectomy on Future Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0232-17-RMB
Record Dates: First submitted 2017-03-29; First posted 2017-04-12 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cyst Ovary
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemostasis with bipolar coagulation (Active Comparator): Patients undergoing laparoscopic ovarian cystectomy with bipolar coagulation hemostasis.
  Interventions: Device: Bipolar coagulation forceps (ETHICON inc.)
- Hemostasis with SURGIFLO (Experimental): Patients undergoing laparoscopic ovarian cystectomy with SURGIFLO hemostasis.
  Interventions: Device: SURGIFLO hemostatic matrix (ETHICON inc.)

INTERVENTIONS:
Device: Bipolar coagulation forceps (ETHICON inc.) — Hemostasis of the base of the ovarian cyst by utilization of a bipolar coagulation device.
  Arms: Hemostasis with bipolar coagulation
Device: SURGIFLO hemostatic matrix (ETHICON inc.) — Hemostasis of the base of the ovarian cyst by utilization of a an absorbable gelatin based matrix known as SURGIFLO.
  Arms: Hemostasis with SURGIFLO

SUMMARY:
Patients undergoing elective laparoscopic ovarian cystectomy will be recruited and randomly divided into 2 groups according to intervention technique-half will be allocated to the bipolar coagulation group and half to the SURGIFLO group.

Patients will be assessed both pre-operatively and 6 months post-operatively by blood tests including follicle stimulating hormone (FSH), lutenizing hormone (LH), Estrogen (E2), Progesterone and anti-mullerian hormone (AMH) levels, and sonographic evaluation of ovarian volume and antral follicle count.

DETAILED DESCRIPTION:
Patients undergoing elective laparoscopic ovarian cystectomy will be recruited after signing an informed consent, and randomly divided into 2 groups according to intervention technique-half will be allocated to the bipolar coagulation group and half to the SURGIFLO group.

Patients will be assessed both pre-operatively and 6 months post-operatively by blood tests including FSH, LH, E2, Progesterone and AMH levels, and sonographic evaluation of ovarian volume and antral follicle count.

Antral follicle count will be performed on the cyst post-surgery using light microscopy. The difference in hormone levels, especially AMH reflects the damage done during surgery to the ovarian reserve. Sonographic signs including a decrease in ovarian volume and antral follicle count also reflect the damage done during surgery to the ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with benign ovarian cysts that are interested in future fertility ages 18-44.

Exclusion Criteria:

* Female patients with malignant ovarian cysts/masses.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients with operable ovarian cysts with clear indication for surgery.
Enrollment: 127 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Decline in ovarian reserve. | Up to 6 months.
  Decline rate of AMH levels before and 6 months after surgery.

SECONDARY OUTCOMES:
Sonographic decline in ovarian volume | Up to 6 months
  Decline rate of ovarian volume before and 6 months after surgery.
Sonographic decline in ovarian antral follicle count | Up to 6 months
  Decline rate of ovarian antral follicle count before and 6 months after surgery.
Changes in FSH levels | Up to 6 months.
  Changes in FSH levels before and 6 months after surgery.
Changes in LH levels | Up to 6 months
  Changes in LH levels before and 6 months after surgery.
Changes in Progesterone levels | Up to 6 months
  Changes in Progesterone levels before and 6 months after surgery.
Changes in E2 levels | Up to 6 months
  Changes in E2 levels before and 6 months after surgery.
Number of antral follicles in the cyst removed from the ovary. | Up to 6 months.
  Number of antral follicles in the cyst removed from the ovary as seen utilizing light microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No